CLINICAL TRIAL: NCT07233317
Title: Evaluating the Safety and Effectiveness of a Vascular Interventional Robotic System in Assisting With Percutaneous Coronary Intervention Procedures: A Prospective, Multicenter, Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-2800
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vascular interventional robotic system group (Experimental): Undergoing PCI using the vascular interventional robotic group
  Interventions: Device: vascular interventional robotic system
- human operator group (Other): Undergoing PCI with human operators
  Interventions: Device: human operator

INTERVENTIONS:
Device: vascular interventional robotic system — Patients all undergoing PCI with vascular interventional robotic system
  Arms: vascular interventional robotic system group
Device: human operator — Patients undergoing PCI by human operators
  Arms: human operator group

SUMMARY:
The goal of this clinical trial is to verify the safety and effectiveness of the vascular interventional robotic system developed and manufactured by Beijing Zhongke Hongtai Medical Technology Co., Ltd. in assisting percutaneous coronary intervention procedures in patients with coronary artery disease. The main question it aims to answer is:

1. Whether the PCI-assisted procedure was clinically successful and technically successful?
2. Will the PCI-assisted procedure can reduce procedure time, PCI time, and radiation exposure for both operators and patients?? Researchers will compare the vascular interventional robotic system with human operators to see if using the vascular interventional robotic system in PCI procedure is effective and safe.

Participants will undergo percutaneous coronary interventions with the vascular interventional robotic system or human operator based on the randomization results. Then all participants will receive a 1-month follow up to evaluate the primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1.18 years ≤ Age ≤ 80 years; 2.Presence of clinical indications for PCI and requiring PCI treatment; 3.The subject or their legal guardian is able to understand the trial objectives, voluntarily signs the informed consent form, and is willing to comply with follow-up procedures.

4.Visual estimation of target lesion diameter stenosis ≥70% (or ≥50% with clinical evidence of myocardial ischemia); 5.2.25 mm ≤ Visual reference vessel diameter ≤ 4.0 mm; 6.The target lesion can be fully covered by a single stent, with at least 2.0 mm of normal vessel segment at the proximal and distal edges of the lesion; 7.Number of target vessels requiring treatment ≤ 2; one target lesion treated with one stent; staged treatment of the target lesion is not allowed.

Exclusion Criteria:

1. Underwent other PCI within 72 hours before the PCI procedure.
2. Underwent PCI within 30 days before the PCI procedure and experienced a Major Adverse Cardiovascular Event (MACE).
3. Experienced acute Myocardial Infarction (MI) within one week before the PCI procedure.
4. Experienced cardiogenic shock within 48 hours before the PCI procedure.
5. Had a stroke within 30 days before the PCI procedure.
6. Subjects with active peptic ulcer or upper gastrointestinal bleeding within 6 months before the PCI procedure.
7. Severe heart failure (NYHA Class IV).
8. Pregnant and lactating women, or women planning to become pregnant during the clinical trial period.
9. Known allergy to aspirin, heparin, clopidogrel, contrast agents, metal materials, etc.
10. Patients with acute or chronic kidney disease (e.g., serum creatinine >2.5 mg/dL or >221 µmol/L) or on dialysis.
11. Subjects with a history of major bleeding or coagulation disorders within the past 6 months.
12. Subjects currently participating in another clinical study that has not completed the entire follow-up period.
13. The investigator determines that the patient has other conditions unsuitable for PCI assisted by the vascular interventional robotic system.
14. Requiring other treatment modalities (such as rotational atherectomy or laser therapy) in addition to balloon angioplasty and stent angioplasty.
15. Presence of more than two lesions in a single vessel requiring simultaneous treatment.
16. Presence of visible thrombus.
17. The target lesion is located in the left main coronary artery.
18. Severely tortuous lesions, severely calcified lesions, or other complex vascular conditions deemed by the investigator as unsuitable for PCI assisted by the vascular interventional robotic system.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Success Rate | Immediately after PCI
Technical Success Rate | Immediately after PCI

SECONDARY OUTCOMES:
Total procedure time | Immediately after PCI
PCI time | Immediately after PCI
Rate of Successful Guiding Catheter Manipulation | Immediately after PCI
Patient Radiation Exposure | Immediately after PCI
Radiation Exposure to Operators and Assistant Physicians | Immediately after PCI
Contrast Agent Volume | Immediately after PCI
Product Performance Evaluation | Immediately after PCI
Incidence of Major Adverse Cardiovascular Events (MACE) | Immediately after PCI and 1 month after PCI
Incidence of Adverse Events and Serious Adverse Events | Immediately after PCI and 1 month after PCI
Incidence of Device Deficiencies | Immediately after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Xicheng District, China

IPD SHARING:
Plan to Share IPD: No
All IPD will not be shared for consideration of personal privacy